CLINICAL TRIAL: NCT02894125
Title: Evaluation of the Effectiveness of a SPA Therapy to "Neyrac-les-Bains" to the Old Subject (60-80 Years Old) With a Chronic Low Back Pain.
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-275
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic Low Back Pain; Old subject; SPA Therapy; Pain; Function; Expectations; Fears
MeSH Terms: conditions — Pain

GROUPS / COHORTS (1):
- old subject
  Interventions: Other: SPA Therapy

INTERVENTIONS:
Other: SPA Therapy

SUMMARY:
Low back pain is considered to be chronic if it has been present for longer than three months.

This pathology is extremely frequent with an annual incidence between 5 in 10 % of the general population. Thus she is frequently met in general medicine, in particular to the ageing subject. It is the 2nd motive for consultation.

The Chronic Low Back Pain is a mild pathology the forecast of which is in the favorable great majority of the cases but she pulled a socioeconomic cost mattering with a poly-consumption of care, in private individuals.

The primary objective of this study is to determine the impact of a 3 months SPA Therapy on the Chronic Low Back Pain in older adults (from 60 to 80 years old) realizing a SPA Therapy of 3 weeks to "Neyrac-les-Bains".

DETAILED DESCRIPTION:
Realization of the protocol :

1. Selection of the patients (realized during the consultation of programming in the beginning of the SPA Therapy). They are 2 thermal doctors of "Neyrac-les-Bains" (1 general practitioner with formation of thermal medicine and a rheumatologist) which include the eligible patients in this study during the visit of the beginning of SPA Therapy.
2. They will put back to the patients the Inform Consent Form, the Form of non-opposition and the 1st questionnaire (J0). The nurse of the SPA Therapy will be at their disposal to help them to fill the questionnaire if need.

An urn will be arranged in the entrance hall of Neyrac- les-Bains to get back the filled questionnaires (J0 and J21).

Patients will follow the conventional SPA Therapy of 3 weeks without a specific changes or modification of the care provided.

Feedback :

Assessments conducted by the using of self - questionnaires:

* Delivered in the issue of the visit of inclusion and at the end of the Spa Therapy ;
* Sent by mail at 3 and 6 months

The expectations and fears will be evaluated by means of individual interview or focus groups. To avoid the biases bound to the questionnaire, the patients questioned in qualitative are different from patients receiving the questionnaire (not over the same period of SPA Therapy).

ELIGIBILITY:
Inclusion Criteria:

* - Both sexes
* 60-80 years old
* Realizing a SPA Therapy of 3 weeks.
* Presenting a mechanical pain of the rachis lumbar vertebra > 3 months
* Possible irradiation up to the knee (cruralgia / sciatalgie truncated)
* Cooperation and understanding allowing to conform in a strict way to the conditions planned by the study
* Acceptance to participate in the study (non-opposition)

Exclusion Criteria:

* - < 60-year-old patients or > 80 years
* Inflammatory, tumoral, traumatic or infectious rheumatism
* Surgery of the back
* SPA Therapy dating less than 6 months
* Evolutionary slipped disc
* Disorders(confusions) of the concentration or the compression of the written or oral French language making impossible the realization of the study
* The pain estimated by the digital scale = 0 in the inclusion

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: old subjects with a chronic low back pain
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pain's estimation by the digital scale | at 3 months

SECONDARY OUTCOMES:
functional incapacity by means of the questionnaire "Oswestry Disability index" | at 0 days, 21 days, 3 months and 6 months
personal efficacy by means of the French questionnaire ASES "Arthritis Self Efficacy Scale" | at 0 day , 21 days, 3 months, 6 months
fears and the faiths with the FABQ (physical dimension only) | at 0 day , 21 days, 3 months, 6 months
consumption of analgesic estimated by a standardized collection | at 21 days, 3 months, 6 months
expectations and fears by means of individual interview or focus groups by means of the quantitative questionnaire for qualitative analysis. | at 0 day

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte ESCHALIER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Rudy TE, Weiner DK, Lieber SJ, Slaboda J, Boston RJ. The impact of chronic low back pain on older adults: a comparative study of patients and controls. Pain. 2007 Oct;131(3):293-301. doi: 10.1016/j.pain.2007.01.012. Epub 2007 Feb 20. PMID 17317008
- [Background] Forestier R, Desfour H, Tessier JM, Francon A, Foote AM, Genty C, Rolland C, Roques CF, Bosson JL. Spa therapy in the treatment of knee osteoarthritis: a large randomised multicentre trial. Ann Rheum Dis. 2010 Apr;69(4):660-5. doi: 10.1136/ard.2009.113209. Epub 2009 Sep 3. PMID 19734131
- [Background] Pittler MH, Karagulle MZ, Karagulle M, Ernst E. Spa therapy and balneotherapy for treating low back pain: meta-analysis of randomized trials. Rheumatology (Oxford). 2006 Jul;45(7):880-4. doi: 10.1093/rheumatology/kel018. Epub 2006 Jan 31. PMID 16449365
- [Background] Koes BW, van Tulder MW, Thomas S. Diagnosis and treatment of low back pain. BMJ. 2006 Jun 17;332(7555):1430-4. doi: 10.1136/bmj.332.7555.1430. No abstract available. PMID 16777886
- [Background] Loney PL, Stratford PW. The prevalence of low back pain in adults: a methodological review of the literature. Phys Ther. 1999 Apr;79(4):384-96. PMID 10201544
- [Derived] Raud B, Lanhers C, Crouzet C, Eschalier B, Bougeard F, Goldstein A, Pereira B, Coudeyre E. Identification of Responders to Balneotherapy among Adults over 60 Years of Age with Chronic Low Back Pain: A Pilot Study with Trajectory Model Analysis. Int J Environ Res Public Health. 2022 Nov 8;19(22):14669. doi: 10.3390/ijerph192214669. PMID 36429387